CLINICAL TRIAL: NCT02554734
Title: Pharmacokinetics of Levodopa After Repeated Doses of Carbidopa, ODM-104 and Levodopa: an Open, Randomised Study With Crossover Design in Healthy Males and Females
Brief Title: Pharmacokinetic Study in Healthy Volunteers
Acronym: NOCOFPK2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3112003
Record Dates: First submitted 2015-06-10; First posted 2015-09-18 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination; entacapone; Stalevo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levodopa standard carbidopa (Experimental): Levodopa, carbidopa, ODM-104
  Interventions: Drug: levodopa, carbidopa, ODM-104
- Levodopa modified carbidopa (Experimental): Levodopa, carbidopa, ODM-104
  Interventions: Drug: levodopa, carbidopa, ODM-104
- Stalevo (Active Comparator): Levodopa, carbidopa, entacapone
  Interventions: Drug: levodopa, carbidopa, entacapone

INTERVENTIONS:
Drug: levodopa, carbidopa, ODM-104
  Other Names: Sinemet
  Arms: Levodopa modified carbidopa; Levodopa standard carbidopa
Drug: levodopa, carbidopa, entacapone
  Other Names: Stalevo
  Arms: Stalevo

SUMMARY:
Phase I open, randomized cross-over pharmacokinetic study.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetics of levodopa, carbidopa, 3-OMD and ODM-104 after repeated doses of levodopa, carbidopa and ODM-104: an open, randomized, multicenter study with crossover design in healthy males and females.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained
* Good general health ascertained by detailed medical history and physical examinations
* Finnish speaking males and females 18-65 years of age
* Normal weight defined as body mass index (BMI) 19-30 kg/m2 (BMI=weight/height m2)
* Weight at least 55 kg
* Regular intestinal transit (no recent history of recurrent constipation, diarrhea, or other intestinal problems, and no history of major gastrointestinal surgery)
* Sexually active study subjects, unless surgically sterile must adhere to a proper form of contraception (hormonal contraception or intrauterine device on female partner, and an additional barrier method used at least by one of the partners) from the first study treatment administration until 3 months after the end-of-study visit

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease or cancer (except local non-melanoma skin cancer) within the previous 2 years.
* Family history (parents, siblings) of clinically significant cardiac conduction disease.
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, paracetamol for occasional pain is allowed. Hormonal contraception and hormone replacement therapy are allowed.
* Intake of any medication that could affect the outcome of the study.
* Any clinically significant abnormal laboratory value or physical finding (including ECG and vital signs) that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject if he/she takes part in the study.
* Known hypersensitivity to the active substances or the excipients of the drugs.
* Pregnant or lactating females.
* History of vasovagal collapses or vagal reactions with unexplained reason within the previous 2 years or a tendency for vasovagal reactions during blood sampling.
* HR < 40 bpm or > 90 bpm in the supine position after 10 min rest at the screening visit.
* At the screening visit:

systolic BP < 90 mmHg or > 150 mmHg in the supine position after 10 min rest diastolic BP < 50 mmHg or > 90 mmHg in the supine position after 10 min rest

* History of anaphylactic/anaphylactoid reactions.
* Strong tendency to motion sickness.
* Recent or current (suspected) drug abuse.
* Recent or current alcohol abuse; regular drinking of more than 21 units per week (males) or 16 units per week (females) (1 unit = 4 cl spirits or equivalent).
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study (from the screening visit to the end-of-study visit).

Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from using caffeine containing beverages 24 h before the first levodopa administration on the PK day (day 7) until collection of the 24 h PK sample in the morning of day 8.

* Blood donation or loss of a significant amount of blood within 90 days before the first study treatment administration.
* Participation in an investigational drug study or administration of an investigational drug within 90 days before the first study treatment administration.
* Veins unsuitable for repeated venipuncture or cannulation.
* Predictable poor compliance or inability to communicate well with the study centre personnel.
* Inability to participate in all treatment periods.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Levodopa Peak Plasma Concentration (Cmax) and fluctuation of levodopa Cmax/Cmin, tau | Blood samples collected frequently on day 7 for 24 hours.
  Explore the Cmax of levodopa and fluctuation of levodopa Cmax/Cmin, tau

SECONDARY OUTCOMES:
Carbidopa Peak Plasma Concentration (Cmax) | Blood samples collected frequently on day 7 for 24 hours.
  Explore Cmax of carbidopa
3-OMD Peak Plasma Concentration (Cmax) | Blood samples collected frequently on day 7 for 24 hours.
  Explore Cmax of 3-OMD
Levodopa Cmax, tau | Blood samples collected frequently on day 7 for 24 hours.
  Explore Cmax, tau of levodopa
Levodopa Cmin, tau | Blood samples collected frequently on day 7 for 24 hours.
  Explore Cmin, tau of levodopa
Levodopa Area under the plasma concentration versus time curve (AUC) | Blood samples collected frequently on day 7 for 24 hours.
  Explore AUC of levodopa
Carbidopa Area under the plasma concentration versus time curve (AUC) | Blood samples collected frequently on day 7 for 24 hours.
  Explore AUC of carbidopa
3-OMD Area under the plasma concentration versus time curve (AUC) | Blood samples collected frequently on day 7 for 24 hours.
  Explore AUC of 3-OMD
Levodopa Peak-trough fluctuation (PTF) | Blood samples collected frequently on day 7 for 24 hours.
  Explore PTF of levodopa

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, Principal Investigator — Clinical Research Services Turku CRST
Locations (1):
- Clinical Research Services Turku CRST, Turku, Finland